CLINICAL TRIAL: NCT01158807
Title: Cerebral Hemorrhage Risk in Hereditary Hemorrhagic Telangiectasia (RDCRN# 6203, Protocol Version Date 07Jan10)
Brief Title: Cerebral Hemorrhage Risk in Hereditary Hemorrhagic Telangiectasia
Acronym: BVMC6203
Status: Active, not recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: RDCRN# 6203; 1U54NS065705 (NIH)
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Hereditary Hemorrhagic Telangiectasia
Keywords: Hereditary Hemorrhagic Telangiectasia; Cerebral arteriovenous malformations
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Intracranial Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood and/or saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HHT- Brain Arteriovenous Malformation: 1. Definite clinical HHT diagnosis (at least 3 Curacao criteria) or genetic diagnosis of HHT and
  2. Presence of Brain Arteriovenous Malformation
- HHT -NO BAVM: 1. Definite clinical HHT diagnosis (at least 3 Curacao criteria) or genetic diagnosis of HHT

SUMMARY:
This study is one of the three projects of an NIH Rare Disease Clinical Research Consortium. A "consortium" is a group of centres sharing information and resources to perform research. The consortium research focuses on brain blood vessel malformations in three different rare diseases.

The focus of this specific study is on Hemorrhagic Telangiectasia (HHT).

HHT is a condition characterized by blood vessel malformations, called telangiectasia and arteriovenous malformations (AVMs), occurring in the brain, nose, lungs, stomach, bowels and liver. Brain AVMs (BAVMs) in HHT are difficult to study because they are rare, affecting approximately 10% of people with HHT. While other types of BAVMs have been studied in depth, studies in the HHT population have been very small. Here, we propose the first large-scale collaboration by joining with 12 HHT Centers of Excellence in North America to perform a large study of risk factors for bleeding from BAVMs, called intracranial hemorrhage (ICH) in HHT patients.

The current standard of clinical practice across North America, is to screen all HHT patients for BAVMs with magnetic resonance imaging (MRI). If BAVMs are detected, patients are referred to a multidisciplinary neurovascular team for consideration for treatment. Treatment decisions are made on a case by case basis, balancing risks of complications from the BAVM with risks of therapy, but are limited by the few studies available in HHT. We hope that the knowledge we obtain about the risk factors for intracranial bleeding in these patients from this larger study will help us to improve the care of HHT patients.

We plan to study risk factors for rupture of BAVMs, including primarily genetics and imaging characteristics of the BAVMs. Knowledge about risk factors will help in the care and management of HHT patients. This will be achieved through the collection of health information to construct a HHT database, blood sampling and banking (through the National Institute of Neurological Disorders and Stroke [NINDS]), and through genetic analysis at the University of California San Francisco.

DETAILED DESCRIPTION:
4. Study Design and Methods In conjunction with the DMCC, we will construct a relational database and web-based data collection instrument; see Table 1 showing the sites that will contribute to this effort. Data will include demographics, symptomology, cerebral angioarchitecture, other organ involvement and HHT gene mutation results.

The database will be used to serve Aim 2 and Aim 3 but will also serve as a platform to foster further HHT research. The recruitment of HHT BAVM cases will be emphasized by use of a 3:1 ratio for enrolling non-BAVM to BAVM HHT cases, i.e., for each brain AVM recruited, 3 patients without a brain AVM will be recruited. This will provide the largest RDCRN 6203 Cerebral Hemorrhage Risk in single sample available that will also have centralized expert neuroradiological adjudication of the brain phenotype.

The study design is detailed, by aim, in Section 6. The data to be collected is detailed in Sections 4.5 and 4.5.1 and the study schedule is detailed in Section 4.6.

4.1. Study Population: The study population will include patients with HHT, with inclusion and exclusion criteria as detailed in section 4.3. Cases will be recruited from two sources: (a) the network of HHT Centers of Excellence (Table 1); and (b) patients who contact study personnel or the HHT Foundation International after learning about the study through the HHT Foundation International social networks, the RDCRN public website, friends, physicians, relatives, etc.

Inclusion and exclusion criteria are detailed in section 4.3. 4.2. Case Ascertainment and Enrollment As shown in Table 2, we estimate conservatively that 875 cases will be available for recruitment over five years. Cases will be derived from two sources. First, we will recruit from the HHT Centers of Excellence cases that are currently being followed and new cases as they pass through the individual clinics. Ascertainment and enrollment will use IRB approved, HIPAA-compliant procedures. Each center will submit cases using web-based forms. Second, we will recruit new cases through the HHT Foundation. The HHT Foundation has a mailing list of 5646 families; there is approximately 1000 new families added per year. HHT Patients who contact the HHT Foundation with an interest in participating in the study will be directed to the closest participating HHT Center of Excellence. The HHT Foundation will recruit patients who contact the HHT Foundation who are interested in participating in the BAVM arm of the study but who are not affiliated with a participating center or do not wish to visit a center to participate in the study. We will also enroll non-BAVM HHT cases to facilitate long-term involvement of the HHT community in systematic, organized rare disease research. We have structured the database to be scalable to accommodate all types of HHT. Under the supervision of the site PI, each local PI and research staff will identify and obtain informed consent from patients and their clinical information is entered into a master registry. At enrollment, arrangements for a blood specimen will also be made. Approximately 20 ml (about 4 teaspoons) of blood will be drawn (two ACD tubes of 8.5 ml each). If a blood draw is not possible, the UCSF core will provide bar-coded saliva DNA collection kits. Representative standard clinical imaging studies (MR and angiography) of enrolled cases will be provided to Dr. Karel TerBrugge at Toronto Western Hospital for adjudication and coding of angioarchitecture. We have conservatively estimated that we will be able to collect DNA from 500 of the 875 project cases that will be enrolled over the course of the study.

4.3 Patient Selection

Inclusion Criteria:

1. (a) Definite clinical HHT diagnosis (at least 3 Curacao criteria) or genetic diagnosis of HHT Curacao criteria: (a) spontaneous recurrent nosebleeds; (b) mucocutaneous telangiectasia at characteristic sites (lips, oral cavity, fingers or the nose); (c) visceral involvement such as pulmonary, hepatic or CNS BAVM; and (d) an affected first degree relative by same criteria.(65) OR (b) Definite clinical HHT diagnosis (at least 3 Curacao criteria) or genetic diagnosis of HHT Curacao criteria: (a) spontaneous recurrent nosebleeds; (b) mucocutaneous telangiectasia at characteristic sites (lips, oral cavity, fingers or the nose); (c) visceral involvement such as pulmonary, hepatic or CNS BAVM; and (d) an affected first degree relative by same criteria.(65) AND Presence of BAVM For the purpose of the study, we will focus on BAVM that directly shunts blood from arterial to venous circulations without an intervening capillary bed, including Toronto classifications(23) of A-V fistulas, "micro" BAVMs (<1 cm) and 8 "small" (1-3 cm) BAVMs, and if present, larger lesions. We will not include intracranial telangiectasias in isolation.
2. Able to provide informed consent Exclusion Criteria: None 4.4 Recruitment and Informed Consent The prospective HHT population will consist of patients seen for evaluation and treatment of HHT. Health status for all patients will encompass a spectrum of disabilities encountered with the disease processes being studied. The Human Subjects Committee/Institutional Review Board of each clinical center will approve the informed consent form. A copy of the letter of approval from the IRB/REB and a copy of the consent form will be filed with the DMCC before a clinical center will be allowed to initiate enrollment. The informed consent will include the objectives of the study, a description of the screening process, the potential risks and benefits, the cost to the patient, alternatives to participation and liabilities of the particular participating center. All patients who are diagnosed with HHT, regardless of gender, race or ethnicity, are potential candidates for the RDCRC. To the best of our knowledge, there is no race-ethnicity predilection for HHT or sporadic BAVMs.

4.5 Data and Sample Collection Development A detailed table of relevant fields and their data types and ranges were constructed by combining elements that are in use by the HHT community and those fields that are collected in our ongoing study of sporadic BAVM. We used these data tables as a departure point to work with the DMCC in constructing both the relational database for the project as well as the data web entry forms. Database issues are also addressed in the GSAC and AU sections.

All recruited participants will be assigned a Database study ID. The link between patient identifying information and database study ID will only be maintained at the recruiting center. Data will be entered through a web-based system into a central Database developed at the DMCC. Only de-identified information will be entered in the central Database.

4.5.1 Detailed Clinical and Radiographic Information to be Collected Information collected will include both attributes of the systemic manifestations of HHT with a focus on the brain vascular phenotype. Detailed tables of data fields and data web entry forms are available from the Site PI, Project Leader, and DMCC. The Clinical data elements include demographic information as well as specific clinical information about clinical features and complications of BAVMs, as well as other organ AVMs and complications related to HHT. The Neuroradiological elements include information about angiographic features, clinical presentation, complications and treatment of BAVMs. This data will be collect at baseline. Every year after recruitment, , participants will be contacted by the recruiting Center to collect a limited follow-up data set, regarding treatment and complications of BAVMs and mortal status.

The diagnosis of BAVM will be made by referring centers and adjudicated by Dr. TerBrugge based on the submitted imaging studies. All imaging studies will be abstracted under the supervision of the consultant neuroradiologist, Dr. TerBrugge. The imaging source and date of CT, MRI, MR angiography, and any diagnostic cerebral angiography furnish primary descriptors including side, nidus size, anatomic location, "eloquence," feeding arteries, arterial aneurysms, number of lesions, and venous drainage pattern. Additional factors include location, the presence of intra- and extranidal aneurysms, and the presence of venous stenoses, as described in the Writing Group paper. New AVM hemorrhage is bleeding into the brain or its surrounding spaces likely to be associated with AVM (age and location of hemorrhage are also estimated). The time from diagnosis to any new hemorrhage will be used in the survival analyses. We will also record other potential sources of co-morbidity, including hypertension, diabetes mellitus, smoking history, hyperlipidemia, i.e., factors that may non-specifically increase the risk of hemorrhage. Although functional status is not part of the primary aims, we will record Modified Rankin Score (mRS)(66-68) (adapted from the ISAT trial patient questions(69)) coded as : 0 = no symptoms and cope well with life; 1 = few symptoms which do not interfere with everyday life; 2 = symptoms which have changed my life but I am still able to look after myself; 3 = symptoms which significantly changed my life, and I need some help looking after myself; 4 = quite severe symptoms, I need help from other people; 5 = major symptoms which severely handicap me and I need constant attention day and night; deaths are coded as 6.

The mRS will be recorded at least for patient status at the time of BAVM discovery and the last available date. For retrospective cases, these will be estimated using available clinical records; for prospective cases, the last available status during the project period will be assessed. New ICH during follow-up will also be recorded. Working with the DMCC, we will institute a web-based system to facilitate data entry. The main follow-up will be targeted to be completed during the fifth year of the RDCRC project and will include: (a) date and nature of any treatment; (b) any new hemorrhagic events; and (c) modified Rankin score.

4.5.2 Sample Collection, Processing and Banking Each site will arrange to obtain a blood sample from BAVM cases, but we will accommodate banking of samples from HHT patients without BAVM for exploratory analyses. Blood samples will be collected and sent directly to the Coriell/NINDS Human Genetics DNA and Cell Line Repository using their published instructions (http://ccr.coriell.org). Coriell with retain DNA and also release a DNA sample to the study investigators UCSF, where it will be stored as well. The advantages of using Coriell/NINDS are (1) 20 μg of genomic DNA will be made available to the researchers at no additional charge, and (2) lymphocytes will be immortalized, ensuring a durable renewable supply of DNA for future studies. The PI has worked with NINDS/Coriell before; we have sent approximately 100 sporadic brain AVM cases to the NINDS DNA bank.

For cases unable to have blood drawn, we will use commercially available saliva mailing kits (Oragene). The kit is sent by the Study Coordinator with instructions for use, consent form, and a return mailing box with pre-printed postage and shipping label. The specimen will be labeled with a study ID number, and sent directly to UCSF for processing and DNA extraction. We have used these with excellent DNA yields and genotyping results. Such samples would be handled directly by the UCSF Genetics and Statistical Analysis Core (GSAC). The Specimen study ID number will be assigned separately from the Database study ID number. Samples will be retained until all DNA has been used up. If there is sample remaining when the study is complete, the study investigators may use the sample for future research studies into genetic factors of and brain AVMs or other aspects of HHT.

ELIGIBILITY:
Inclusion criteria:

* Definite clinical HHT diagnosis (at least 3 Curacao criteria)or genetic diagnosis of HHT or
* Definite clinical HHT diagnosis (at least 3 Curacao criteria) or genetic diagnosis of HHT and Presence of Brain Arteriovenous Malformation
* Able to provide informed consent

Curacao criteria:

1. spontaneous recurrent nosebleeds;
2. mucocutaneous telangiectasia at characteristic sites (lips, oral cavity or the nose);
3. visceral involvement such as pulmonary, hepatic or CNS BAVM; and (d) an affected first degree relative by same criteria.

Willingness

* Willingness to participate in the study and ability to give informed consent

Exclusion Criteria:

* Patients not complying with Inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HHT individuals with a history of brain arteriovenous malformation. HHT individuals without a history of brain arteriovenous malformation.
Sampling Method: Non-Probability Sample
Enrollment: 2272 (Actual)
Dates: Start 2010-04-08 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Aim 1: The identification of predictors of brain outcomes in HHT patients | Through study completion, an average of 5 years
  This study will investigate predictors of brain outcomes in HHT patients. The investigators hypothesize that the presence of brain arteriovenous malformation (BAVM) in HHT patients versus HHT patients without BAVM and multiplicity of BAVMs will be associated with worsening functional outcome. Therefore, the comprehensive brain outcomes in HHT for future HHT clinical trials will be characterized.

SECONDARY OUTCOMES:
Aim 2: A severe bleeding phenotype in HHT will be defined for clinical trial readiness | Through study completion, an average of 5 years
  The investigators hypothesize that weekly nasal bleeding duration in HHT will predict the need for invasive or life-sustaining therapies. HHT participant reported bleeding duration will be measured longitudinally and correlate with the need for invasive or life-sustaining therapies, as well as with ICH risk from BAVMs and with bleeding in other HHT organ phenotypes.
Aim 3: The genetic predictors and circulating biomarkers of severe bleeding and brain outcomes in HHT will be characterized | Through study completion, an average of 5 years
  The investigators hypothesize that there are shared predictors of severe bleeding from the nose and brain in HHT patients, and that identifying these predictors will allow for selection of "at-risk" patients for clinical trials. Specifically, potential genetic, plasma protein biomarker and circulating miRNA biomarker predictors of bleeding will be evaluated. Markers associated with bleeding will then be tested for association with ICH, and with other brain outcomes and HHT severity phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Faughnan, MD MSc FRCPC, Principal Investigator — Unity Health Toronto
Locations (19):
- United States (14):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - David Geffen School of Medicine at University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - UCHealth Pulmonary Vascular Disease Clinic - Anschutz Medical, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Georgia Regents University, Augusta, Georgia
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - HHT Foundation International, Inc., Monkton, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, NC, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Utah, Salt Lake City, Utah
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - St. Paul's Hospital, University of British Columbia, Vancouver, British Columbia
  - St. Michael's Hospital, Toronto, Ontario
  - Hospital for Sick Children, Toronto, Ontario
- St. Antonius Hospital, Nieuwegein, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: This is the Rare Diseases Clinical Research Networkweb site which lists the BVMC 6203 HHT study — https://www.rarediseasesnetwork.org/cms/bvmc/Get-Involved/Studies/6203-HHT